CLINICAL TRIAL: NCT01052090
Title: Safety and Efficacy Study in Non-Responder Hepatitis C Genotype 1 Patients With PHN121
Brief Title: Safety and Efficacy Study in Hepatitis C Patients With PHN121
Acronym: ENCHAMP
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PH-CP015
Record Dates: First submitted 2010-01-17; First posted 2010-01-20 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2010-01

CONDITIONS: Hepatitis C Virus Infection
Keywords: HCV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Drug: PHN121

INTERVENTIONS:
Drug: PHN121 — a size 0 hard gel capsule containing 323.6 mg active ingredient, a complex mixture prepared from 5 commonly practiced botanical traditional Chinese medicines

SUMMARY:
To evaluate the safety, tolerability and efficacy of escalating dose of PHN121 when administered orally in non-responder hepatitis C genotype 1 patients

DETAILED DESCRIPTION:
This is a Phase I/II, open-label, multicenter (2 centers), dose-escalation, multidose study in non-responder hepatitis C genotype 1 patients. Three escalating dose levels will be evaluated. Each cohort of 6 subjects will enroll sequentially. Each cohort will be administered PHN121 orally daily for 12 weeks. Subjects will be requested to return on Week 2, Week 4, Week 6, and Week 9 for evaluation and medication. Subjects will also be asked to return for follow-up evaluation for adverse events on Week 12 and Week 16.

Three doses are planned and include: 2.91, 4.85, and 7.77 g/day. Subjects will be assigned to a dose level in the order of study entry. Initially, 6 subjects will be enrolled at each dose level; up to 8 subjects may be assigned to each dose level, depending upon dose-limiting toxicities (DLTs) seen.

Six subjects will be started on treatment with dose level 1. After the sixth subject completes 84 days of treatment, if no dose-limiting toxicity occurs, then the next group of 6 subjects will be treated at the next higher dose regimen. If 1 of the 6 initial subjects experiences a DLT, the cohort of subjects will be expanded to 8 subjects. If fewer than two DLTs occur in 8 subjects, then the next higher dose group will be initiated. If 2 of the 6 initial subjects or 3 or more (of a cohort of up to 8) subjects experience DLTs, no further dose escalations will occur; the study will be discontinued and the MTD will have been exceeded.

No subject may participate in more than 1 cohort.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking adult subjects age 20 years or above, male or female
* Non-Responder HCV patient who failed to achieve sustained viral response (SVR), either do not respond or relapse, to prior 24-week interferon based therapy
* Any antiviral agent discontinued at least 4 weeks before the screening visit.
* Presence of anti-HCV in serum
* Serum and PCR positive for HCV-RNA*1 (Genotype 1)
* Elevated ALT (> 1.3 x upper limit of normal) during last 6 months and (1.3 x to 10 x upper limit of normal) during the screening phase
* No evidence showing liver cirrhosis or hepatocellular carcinoma*2
* Hematological, biochemical and serologic criteria at the screening phase is within normal limits (WNL):

  * Hemoglobin values of > 12gm/dl for females and > 13gm/dl for males
  * WBC > 3,000/mm3
  * Neutrophil > 1,500/mm3
  * Platelets count > 90,000/mm3
  * Normal PT (INR< 1.2)
  * Total bilirubin < 2 mg/dl
  * Albumin, WNL
  * Serum creatinine, WNL
* Written informed consent

Exclusion Criteria:

* Has evidence of significant renal, cardiovascular, hematopoetic, neurological, pulmonary or gastrointestinal pathology, or any other medical reason or disease that might interfere with the study objectives, as determined by the investigator
* Has participated in other investigational trials within 28 days prior to study enrollment
* Has taken botanical medications*3 within 28 days prior to study enrollment
* Has an surgery within 28 days prior to study enrollment
* Has been diagnosed with any other cause for the liver disease other than chronic hepatitis C including the following conditions:

  * Co-infection with HBV
  * Hemochromatosis
  * Alpha-1 antitrypsin deficiency
  * Wilson's disease
  * Autoimmune hepatitis
  * Alcoholic liver disease
  * Drug-related liver disease
  * Other liver disease that was considered by the principal investigator
* Has been test positive for HIV
* Has been diagnosed with poor-controlled Diabetes Mellitus (HbA1C > 9.0%)
* Active alcohol abuse of daily intake > 30 g for male and > 20 g for female within the previous 1 year
* Active substance abuse, such as inhaled or injection drugs within the previous 1 year *4
* Female subjects of child bearing potential who are pregnant, nursing, do not agree to practice effective birth control during the time period from 14 days before administration of study drug to 28 days after administration of study drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Safety: Safety assessments will include ALT, aspartate aminotransferase (AST), other clinical laboratory tests, HCV RNA quantitation, vital signs, physical examinations, concomitant medications, and adverse events (AEs). | 12-week treatment; 4-week safety followup

SECONDARY OUTCOMES:
Efficacy: Efficacy will be assessed by evaluating the plasma concentrations of ALT and viral load through calculating the percent change from Baseline on a per-subject and by-cohort basis, normalizing to the baseline measurement. | 12-week treatment; 4-week safety followup

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Long Chuang, M.D., Ph.D., Principal Investigator — Kaohsiung Municipal United Hospital; Ming-Lung Yu, M.D., Ph.D., Principal Investigator — Kaohsiung Municipal United Hospital; Chia-Yen Dai, M.D., M.S., Principal Investigator — Kaohsiung Municipal United Hospital
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - PhytoHealth, Taipei

REFERENCES:
- [Background] Dai CY, Chuang WL, Huang JF, Hsieh MY, Yu ML. Rapid virological response in hepatitis C virus genotype 1 and early ribavirin exposure. Hepatology. 2008 Aug;48(2):692-3; author reply 693-4. doi: 10.1002/hep.22409. No abstract available. PMID 18666250
- [Background] Huang JF, Dai CY, Lin YY, Yu ML, Liu SF, Lin IL, Hsieh MY, Lee LP, Lin ZY, Chen SC, Hsieh MY, Chang WY, Chuang WL. Performance characteristics of a real-time RT-PCR assay for quantification of hepatitis C virus RNA in patients with genotype 1 and 2 infections. Clin Chem Lab Med. 2008;46(4):475-80. doi: 10.1515/CCLM.2008.082. PMID 18605932